CLINICAL TRIAL: NCT00192023
Title: An Italian Randomised, Double-blind Placebo Controlled Study of the Efficacy of Atomoxetine Hydrochloride in the Treatment of Children and Adolescents With Attention-Deficit/Hyperactivity Disorder and Comorbid Oppositional Defiant Disorder
Brief Title: An Italian Study of the Efficacy of Atomoxetine in the Treatment of Children and Adolescents With Attention-Deficit/Hyperactivity Disorder (ADHD) and Comorbid Oppositional Defiant Disorder (ODD).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chielf Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8856; B4Z-IT-LYCY (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2010-01-18 (Estimated); Last update posted 2010-01-18 (Estimated); Status verified 2009-12

CONDITIONS: Attention Deficit Hyperactivity Disorder; Oppositional Defiant Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Oppositional Defiant Disorder | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atomoxetine (Experimental): atomoxetine 0.5 milligrams per kilogram per day (mg/kg/day) daily (QD), by mouth (PO) for 1 week, 1.2 mg/kg/day QD, PO for 7 weeks, then 1.2 - 1.4 mg/kg/day QD, PO for up to 1.5 years or until atomoxetine receives marketing approval.
  Interventions: Drug: atomoxetine 0.5 mg/kg/day; Drug: atomoxetine 1.2 mg/kg/day; Drug: atomoxetine 1.2-1.4 mg/kg/day
- Placebo (Placebo Comparator): placebo, daily (QD), by mouth (PO) for 8 weeks, then possibility to switch to atomoxetine at 0.5 mg/kg/day QD, PO for 1 week, then to 1.2 - 1.4 mg/kg/day QD, PO for up to 1.5 years or until atomoxetine receives marketing approval.
  Interventions: Drug: atomoxetine 0.5 mg/kg/day; Drug: placebo; Drug: atomoxetine 1.2-1.4 mg/kg/day

INTERVENTIONS:
Drug: atomoxetine 0.5 mg/kg/day — atomoxetine 0.5 milligrams per kilogram per day (mg/kg/day) daily (QD), by mouth (PO)
  Other Names: LY139603; Strattera
Drug: placebo
  Arms: Placebo
Drug: atomoxetine 1.2 mg/kg/day — atomoxetine 1.2 mg/kg/day QD, PO
  Other Names: LY139603; Strattera
  Arms: Atomoxetine
Drug: atomoxetine 1.2-1.4 mg/kg/day — atomoxetine 1.2 - 1.4 mg/kg/day QD, PO
  Other Names: LY139603; Strattera

SUMMARY:
The study is a phase IIIb multicentre, randomised, placebo controlled, trial in paediatric patients with Attention-Deficit/Hyperactivity (ADHD) and Oppositional Defiant Disorder (ODD). The primary aim of the study is to evaluate the efficacy of atomoxetine in improving ADHD and ODD symptoms in patients non responders to a previous psychological intervention with parent support. Moreover, the potential role of atomoxetine in treating other psychiatric comorbid conditions associated with ADHD and ODD will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Child or adolescent patients, male or female outpatients, who are at least 6 years of age, but must not yet have reached their 16th birthday prior to Visit 1, when informed consent is obtained.
* Patients must meet Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) diagnostic criteria for ADHD (any subtype) and ODD and score at least 1.5 standard deviations above the age norm for their diagnostic subtype using published norms for the Swanson, Nolan and Pelham Questionnaire: Attention-Deficit/Hyperactivity Disorder (SNAP-IV ADHD) Subscale score at both Visit 1 and 2.
* They must also have a SNAP-IV ODD subscale score of at least 15 at both Visit 1 and Visit 2.
* Other comorbid conditions, are allowed but the diagnosis of ADHD and ODD must be the patient's primary diagnosis.
* Patients must be of normal intelligence in the judgment of the investigator (that is, without a general impairment of intelligence and likely, in the investigator's judgement, to achieve a score of greater than or equal to 70 on an Intelligence Quotient (IQ) test). The administration of a formal IQ test is not an entry requirement for the study. Specific learning disabilities are not considered general impairment of intelligence.

Exclusion Criteria:

* Patients who weigh less than 20 kilograms (kg) at study entry (Visit 1).
* Patients who have a documented history of Bipolar I or II disorder, any history of psychosis or pervasive development disorder.
* Patients with a history of any seizure disorder (other than febrile seizures) or patients who have taken (or are currently taking) anticonvulsants for seizure control are not eligible to participate.
* Patients at serious suicidal risk as assessed by the investigator.
* Patients who, in the investigator's judgment, are likely to need psychotropic medications apart from the drug under the study, including health-food supplements that the investigator feels have central nervous system activity (for example, St. John's Wort, melatonin).

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 139 (Actual)
Dates: Start 2004-10; Primary Completion 2006-08 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST ), Study Director — Eli Lilly and Company
Locations (12):
- Italy (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Alessandria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Bari
  - For additional Information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Cagliari
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Genova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Messina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Napoli
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Padua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Pavia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Pisa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Roma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., S. Vito Tagliamento
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Venezia

REFERENCES:
- [Derived] Bangs ME, Wietecha LA, Wang S, Buchanan AS, Kelsey DK. Meta-analysis of suicide-related behavior or ideation in child, adolescent, and adult patients treated with atomoxetine. J Child Adolesc Psychopharmacol. 2014 Oct;24(8):426-34. doi: 10.1089/cap.2014.0005. Epub 2014 Jul 14. PMID 25019647
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study Period I=Screening. Study Period II=Standardized behavioral management program for parents (156 entered, 17 discontinued). Study Period III=Double-Blind (randomization). Two patients did not have post-baseline values for the primary endpoint and were not included in Baseline or efficacy analyses. Study Period IV=Optional open-label phase.
Groups:
- Atomoxetine: atomoxetine 0.5 mg/kg/day daily (QD), by mouth (PO) for 1 week, 1.2 mg/kg/day QD, PO for 7 weeks, then 1.2 - 1.4 mg/kg/day QD, PO for up to 1.5 years or until atomoxetine received marketing approval.
- Placebo: placebo, daily (QD), by mouth (PO) for 8 weeks, then possibility to switch to atomoxetine at 0.5 mg/kg/day QD, PO for 1 week, then to 1.2 - 1.4 mg/kg/day QD, PO for up to 1.5 years or until atomoxetine received marketing approval.
Period: Period III - Double-Blind
Arm/Group | Atomoxetine | Placebo
Started | 107 | 32
Completed | 100 (6 patients who completed the protocol did not enter optional open-label period.) | 32 (2 patients who completed the protocol did not enter the optional open-label period.)
Not Completed | 7 | 0
Not completed — Adverse Event | 3 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Parent/Caregiver Decision | 2 | 0
Period: Period IV - Optional Open-Label
Arm/Group | Atomoxetine | Placebo
Started | 124 | 0 (Placebo patients received atomoxetine during the optional open-label period.)
Completed | 49 | 0
Not Completed | 75 | 0
Not completed — Adverse Event | 6 | 0
Not completed — Lack of Efficacy | 7 | 0
Not completed — Patient/Caregiver Decision | 46 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Physician Decision | 9 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atomoxetine | Placebo | Total
Number analyzed (Participants) | 105 | 32 | 137
Age Continuous [Mean (Standard Deviation); unit: years] | 9.7 (2.2) | 10.0 (2.4) | 9.8 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 98 | 29 | 127
Region of Enrollment [Number; unit: participants]
  Italy | 105 | 32 | 137
Race/Ethnicity [Number; unit: participants]
  Caucasian | 104 | 29 | 133
  Hispanic | 1 | 3 | 4
Height [Mean (Standard Deviation); unit: centimeters] | 140.1 (15.2) | 141.6 (15.3) | 140.4 (15.1)
Weight [Mean (Standard Deviation); unit: kilograms] | 39.3 (15.8) | 41.4 (14.1) | 39.8 (15.4)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 8 Week Endpoint in Swanson, Nolan and Pelham Questionnaire (SNAP-IV): Attention-Deficit/Hyperactivity Disorder (ADHD) Subscale
Description: Items from the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) criteria for ADHD are included for the two subsets of symptoms: inattention (items #1-#9) and hyperactivity/impulsivity (items #11-#19). The SNAP-IV is based on a 0 (not at all) to 3 (very much) rating scale. Total subscale scores range from 0 to 54.
Time Frame: Visit 8 (baseline) and Visit 14 (8 weeks)
Population: Efficacy Population (All 139 randomized patients with at least a post-baseline value for the primary endpoint, i.e, 105 + 32 = 137 patients in total). Last Observation Carried Forward was applied.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 105 | 32
units on a scale
  Baseline | 42.7 (6.2) | 41.5 (6.9)
  Change to 8 Week Endpoint | -8.1 (9.2) | -2.0 (4.7)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Using an estimate of the common standard deviation of 13 points, the planned sample size will give about 80% power to detect a difference between the groups of 8 points on the SNAP-IV. The sample size was determined using a two-sided test with p=0.05, and assumes that up to 10% of patients will discontinue the study without providing post-baseline efficacy data in Study Period III; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Change to Week 8 Endpoint. Change = Endpoint minus baseline. Model: Change to Week 8=score at Week 8+treatment+site+treatment-by-site interaction. If treatment-by-site interaction isn't significant it will be removed from model

2. Secondary Outcome: Change From Baseline to 8 Week Endpoint in Clinical Global Impressions - Attention-Deficit/Hyperactivity Disorder (ADHD) - Severity
Description: Measures severity of illness at the time of assessment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients.
Time Frame: Visit 8 (baseline) and Visit 14 (8 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 105 | 32
units on a scale
  Baseline | 5.1 (0.8) | 5.1 (0.9)
  Change to 8 Week Endpoint | -0.6 (0.7) | 0.0 (0.5)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Change to 8 Week Endpoint. Change = Endpoint minus baseline. Model: Change to 8 Week Endpoint=Score at 8 weeks+treatment+site

3. Secondary Outcome: Change From Baseline to 8 Week Endpoint in SNAP-IV Oppositional Subscale
Description: Items are included from the DSM-IV criteria for Oppositional Defiant Disorder (items #21-#28). The SNAP-IV is based on a 0 (not at all) to 3 (very much) rating scale. Total subscale scores range from 0 to 24.
Time Frame: Visit 8 (baseline) and Visit 14 (8 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 105 | 32
units on a scale
  Baseline | 17.2 (3.0) | 17.5 (3.8)
  Change to 8 Week Endpoint | -2.7 (4.1) | -0.3 (2.6)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]

4. Secondary Outcome: Change From Baseline to 8 Week Endpoint in Screen for Child Anxiety Related Emotional Disorders (SCARED) Total Score
Description: The scale measures symptoms of DSM-IV linked anxiety disorders in children. Contains 41 items. Individual item scores range from 0 (not true or hardly ever true) to 2 (very true or often true). Therefore, the overall score ranges from 0 to 82. Higher scores are more indicative of greater anxiety.
Time Frame: Visit 8 (baseline) and Visit 14 (8 weeks)
Population: Efficacy Population (All 139 randomized patients with at least a post-baseline value for the primary endpoint, i.e., 105 + 32 = 137 patients in total). Last Observation Carried Forward was applied. Missing data were not imputed, which generates different analysis population sizes for the different endpoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 103 | 32
units on a scale
  Baseline | 20.3 (11.8) | 18.8 (11.5)
  Change to 8 Week Endpoint | -2.1 (7.6) | -1.7 (6.5)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.836, ANCOVA — [p-value comment as in outcome 2, analysis 1]

5. Secondary Outcome: Change From Baseline to 8 Week Endpoint in Children's Depression Rating Scale-Revised
Description: Measures presence and severity of depression. Consists of 17 items scored on a 1-5 or 1-7 scale. A rating of 1 indicates normal, thus the minimum score is 17. The maximum score is 113. In general, scores below 20 indicate an absence of depression; scores of 20 or 30 indicate borderline depression; scores of 40 to 60 indicate moderate depression.
Time Frame: Visit 8 (baseline) and Visit 14 (8 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 105 | 32
units on a scale
  Baseline | 28.0 (8.4) | 26.9 (8.1)
  Change to 8 Week Endpoint | -0.5 (4.4) | -0.1 (5.0)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.870, ANCOVA — [p-value comment as in outcome 2, analysis 1]

6. Secondary Outcome: Change From Baseline to 8 Week Endpoint in Conners' Parent Rating Scale-Revised: Short Form Subscale Scores
Description: A 27-item rating scale (0 [not at all/never] to 3 [very much true/very often]) completed by the parent to assess problem behaviors related to ADHD. Subscales: Oppositional, Cognitive Problems, Hyperactivity, and ADHD Index. Subscale total scores range from 0 to 18 for all subscales except ADHD Index which ranges from 0 to 36.
Time Frame: Visit 8 (baseline) and Visit 14 (8 weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 103 | 32
units on a scale
  Oppositional Baseline | 11.7 (3.8) | 12.2 (3.9)
  Oppositional Change to 8 Week Endpoint | -1.2 (3.9) | 0.8 (2.7)
  Cognitive Problems Baseline | 14.3 (3.1) | 14.2 (3.2)
  Cognitive Problems Change to 8 Week Endpoint | -2.3 (3.8) | 0.2 (2.6)
  Hyperactivity Baseline | 12.0 (3.8) | 12.0 (4.0)
  Hyperactivity Change to 8 Week Endpoint | -2.2 (4.1) | -0.7 (2.6)
  ADHD Index Baseline | 28.2 (4.9) | 28.4 (5.2)
  ADHD Index Change to 8 Week Endpoint | -5.0 (6.7) | -0.1 (3.9)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.002, ANCOVA — P-value for Oppositional Change to 8 Week Endpoint. Change = Endpoint minus baseline. Model: Change to 8 Week Endpoint=Score at 8 weeks+treatment+site
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Cognitive Problems Change to 8 Week Endpoint. Change = Endpoint minus baseline. Model: Change to 8 Week Endpoint=Score at 8 weeks+treatment+site
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.022, ANCOVA — P-value for Hyperactivity Change to 8 Week Endpoint. Change = Endpoint minus baseline. Model: Change to 8 Week Endpoint=Score at 8 weeks+treatment+site
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for ADHD Index Change to 8 Week Endpoint. Change = Endpoint minus baseline. Model: Change to 8 Week Endpoint=Score at 8 weeks+treatment+site

7. Secondary Outcome: Change From Baseline to 8 Week Endpoint in Child Health and Illness Profile - Child Edition (CHIP-CE): Parent Rated Form
Description: Parent-rated assessment of a child's health status and level of functioning. It consists of 76 items. The majority of items assess frequency of activities or feelings using a five-point response format (for example, 'how good is your child at making friends?' 1=never, 5=always). Standard scores (t-value) were established, with all domains and subdomains having a mean score of 50 and standard deviation of 10. Standard scores are expressed in standard deviation units. T-score=[(score-4.2382)*10/0.32835] + 50. Higher scores mean improvement.
Time Frame: Visit 8 (baseline) and Visit 14 (8 weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: standard deviation units
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 97 | 29
standard deviation units
  Baseline | 27.1 (10.4) | 26.9 (11.2)
  Change to 8 Week Endpoint | 3.6 (8.0) | 1.2 (6.6)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.071, ANCOVA — [p-value comment as in outcome 2, analysis 1]

8. Secondary Outcome: Change From Baseline to 8 Week Endpoint in Conners' Teacher Rating Scale-Revised: Short Form Subscale Scores
Description: A 28-item rating scale (0 [not at all/never] to 3 [very much true/very often]) completed by the teacher to assess problem behaviors related to ADHD. Subscale total scores range from 0 to 15 for Oppositional and Cognitive Problems, 0 to 21 for Hyperactivity, and 0 to 36 for ADHD Index.
Time Frame: Visit 8 (baseline) and Visit 14 (8 weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 58 | 18
units on a scale
  Oppositional Baseline | 7.6 (4.3) | 10.8 (3.8)
  Oppositional Change to 8 Week Endpoint | -1.1 (2.9) | 0.1 (2.2)
  Cognitive Problems Baseline | 8.2 (4.3) | 8.5 (3.7)
  Cognitive Problems Change to 8 Week Endpoint | -0.9 (2.5) | 0.0 (1.7)
  Hyperactivity Baseline | 12.8 (5.5) | 16.3 (3.4)
  Hyperactivity Change to 8 Week Endpoint | -2.1 (4.7) | -1.1 (3.0)
  ADHD Index Baseline | 25.3 (8.4) | 29.4 (6.0)
  ADHD Index Change to 8 Week Endpoint | -3.5 (7.1) | -0.9 (3.3)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.002, ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.113, ANCOVA — [p-value comment as in outcome 6, analysis 2]
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.051, ANCOVA — [p-value comment as in outcome 6, analysis 3]
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.061, ANCOVA — [p-value comment as in outcome 6, analysis 4]

9. Other Pre Specified Outcome: Open-Label Phase Serious Adverse Events
Description: Number of participants with serious adverse events during the open-label phase of the trial, which was for 1.5 years or until atomoxetine received marketing approval.
Time Frame: Baseline (Visit 14) though 1.5 years (Visit 20) or until atomoxetine received marketing approval
Population: Number of patients who entered this optional open-label phase. All of the patients were dispensed drug.
Measure: Number; unit: participants
Arm/Group | Atomoxetine
Number analyzed (Participants) | 124
participants
  Vomiting | 1
  Infectious mononucleosis | 1
  Agitation | 1

10. Other Pre Specified Outcome: Open-Label Phase Nonserious Adverse Events
Description: Number of participants with nonserious adverse events during the open-label phase of the trial, which was for 1.5 years or until atomoxetine received marketing approval.
Time Frame: Baseline (Visit 14) though 1.5 years (Visit 20) or until atomoxetine received marketing approval
Population: Number of patients who entered this optional open-label phase. All of the patients were dispensed drug.
Measure: Number; unit: participants
Arm/Group | Atomoxetine
Number analyzed (Participants) | 124
participants
  Abdominal pain | 6
  Nausea | 10
  Vomiting | 11
  Pyrexia | 6
  Influenza | 7
  Weight decreased | 5
  Anorexia | 10
  Decreased appetite | 7
  Headache | 19
  Somnolence | 8
  Agitation | 7
  Insomnia | 4

ADVERSE EVENTS:
Time Frame: The results in this module are serious (there weren't any) and non-serious adverse events during Study Period III. Adverse events during the Open-Label (Period IV) phase are presented as Other Pre-Specified Outcome Measures.
Arm/Group | Atomoxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/107 | 0/32
Other Adverse Events (participants affected / at risk) | 79/107 | 12/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=107) | Placebo (N=32)
Abdominal pain (Gastrointestinal disorders) | 11 (13) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 9 (11) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 4 (6) | 2 (2)
Nausea (Gastrointestinal disorders) | 14 (15) | 0 (0)
Vomiting (Gastrointestinal disorders) | 14 (22) | 1 (1)
Influenza (Infections and infestations) | 9 (9) | 0 (0)
Weight decreased (Investigations) | 6 (6) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 26 (27) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 9 (10) | 0 (0)
Headache (Nervous system disorders) | 18 (22) | 4 (5)
Somnolence (Nervous system disorders) | 18 (19) | 2 (2)
Nervousness (Psychiatric disorders) | 6 (6) | 1 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Due to the open-ended timing of the open-label period (up to 1.5 years or until commercial availability) the efficacy data from the open-label extension phase is not included except for adverse event data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days